CLINICAL TRIAL: NCT03052075
Title: Percent Change in Baseline Bone Mineral Density (BMD) After Parathyroidectomy in Patients With Primary Hyperparathyroidism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA14-0401
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Primary Hyperparathyroidism
Keywords: Primary Hyperparathyroidism; Parathyroidectomy; Bone mineral density; BMD; Data Review
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parathyroidectomy Data Review: The research plan is for a retrospective review to be performed of a prospectively maintained parathyroid database within the Department of Surgical Oncology at the University of Texas MD Anderson Cancer Center.
  Interventions: Other: Retrospective Data Review

INTERVENTIONS:
Other: Retrospective Data Review — Retrospective, uncontrolled pre- and post-test design in a case series of approximately 250 patients who underwent parathyroidectomy at MD Anderson Cancer Center (years 1990 - 2013 ) and had bone density measures recorded at baseline and at one year post-surgery. Data extracted from the surgical oncology database for bone mineral density measures for each patient at multiple sites including the lumbar spine, total hip (right/left), femoral neck (right/left), and distal 1/3 radius. All measures recorded from two time points: presurgical (baseline) and postsurgical (all follow-up available dates beginning at 1 year post-parathyroidectomy).

SUMMARY:
The primary objective of this study is to estimate the percent change in baseline bone mineral density (BMD) starting at one year after parathyroidectomy and all the following available dates in patients presenting with primary hyperparathyroidism. The secondary objective is to identify patient factors associated with change in BMD.

DETAILED DESCRIPTION:
The research plan is for a retrospective review to be performed of a prospectively maintained parathyroid database within the Department of Surgical Oncology at the University of Texas MD Anderson Cancer Center. The patient cohort for this study consists of all patients with primary hyperparathyroidism who underwent parathyroidectomy and also had pre- and post-operative DEXA studies performed. The database will be reviewed to obtain patient and disease characteristics, laboratory values, DEXA imaging results, and surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. The patient cohort for this study consists of all patients within the prospectively maintained parathyroid database within the Department of Surgical Oncology at the University of Texas MD Anderson Cancer Center.
2. Patients with a diagnosis of primary hyperparathyroidism who underwent parathyroidectomy during the period of September 27, 1990 to December 31, 2013 were considered.
3. All patients who had a preoperative and one year post-operative DEXA study over the time period will be included.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient cohort for this study consists of all patients with primary hyperparathyroidism who underwent parathyroidectomy and also had pre- and post-operative DEXA studies performed at MD Anderson Cancer Center.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-09-03 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Bone Mineral Density | Baseline to at least one year after parathyroidectomy
  Data from the pre- and post-tests plotted and correlations assessed using the Pearson or Spearman rank correlation coefficient. Differences in pre- and post-operative bone mineral density measures at each site tested using a paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org